CLINICAL TRIAL: NCT04693507
Title: An Adaptive Phase 2, Open-Label, Multicentre Study Investigating the Pharmacokinetics, Pharmacodynamics, Efficacy and Safety of Teverelix Trifluoroacetate, a GnRH Antagonist, in Participants With Advanced Prostate Cancer
Brief Title: Teverelix Evaluated in Advanced Prostate Cancer
Acronym: TEACh
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antev Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANT-1111-02
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-01

CONDITIONS: Prostatic Adenoma
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Adaptive design - enrollment will open in Group 1 (6-weekly dosing regimen). Only if Group 1 dosing regimen is unsuccessful will enrollment open in Group 2 (4-weekly dosing regimen)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teverelix TFA 120 mg 6-weekly (Experimental): Participants receive teverelix TFA loading dose on Day 0 (120 mg SC + 120 mg IM) and teverelix TFA maintenance doses of 120 mg SC at week 6 and 6-weekly thereafter up to week 24
  Interventions: Drug: teverelix TFA 120 mg
- Teverelix TFA 180 mg 6-weekly (Experimental): Participants receive teverelix TFA loading dose on Day 0 (180 mg SC + 180 mg IM) and teverelix TFA maintenance doses of 180 mg SC at week 6 and 6-weekly thereafter up to week 24
  Interventions: Drug: teverelix TFA 180 mg

INTERVENTIONS:
Drug: teverelix TFA 120 mg — Teverelix TFA 240 mg Day 0 and 120 mg every 6 weeks from week 6 to week 24
  Arms: Teverelix TFA 120 mg 6-weekly
Drug: teverelix TFA 180 mg — Teverelix TFA 360 mg Day 0 and 180 mg every 6 weeks from week 6 to week 24
  Arms: Teverelix TFA 180 mg 6-weekly

SUMMARY:
The purpose of this study is to assess the safety and efficacy of teverelix TFA in the treatment of advanced prostate cancer

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo an up to 7 day screening period to determine eligibility for study entry. On Day 0, patients who meet the eligibility requirements will be enrolled in an open-label manner and will receive a loading dose of teverelix TFA (one subcutaneous (SC) injection in the abdomen and one intramuscular (IM) injection in the buttock). Patients will then receive maintenance doses of teverelix TFA (one SC injection in the abdomen) at 4- or 6-weekly intervals up to week 24. The patients will return for a final assessment 4 weeks after their last maintenance dose injection.

The initial dosing regimen to be tested (Group 1) is:

Loading Dose = 120 mg teverelix TFA SC + 120 mg teverelix TFA IM Maintenance Dose = 120 mg teverelix TFA SC every 6 weeks

If this dosing regimen is unsuccessful (more than 2 (of 20) patients fail treatment) then recruitment to Group 1 will end and enrollment in Group 2 will open.

The dosing regimen that may be tested (Group 2) is:

Loading Dose = 180 mg teverelix TFA SC + 180 mg teverelix TFA IM Maintenance Dose = 180 mg teverelix TFA SC every 6 weeks

If this dosing regimen is unsuccessful (more than 6 (of 60) patients fail treatment) then recruitment to Group 2 will end and the study will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* Is male, aged ≤80 years (≥18 years) at the beginning of the treatment period (Day 0)
* Has histologically proven advanced adenocarcinoma of the prostate (metastatic or non metastatic hormone-sensitive non curative), suitable for ADT
* Is treatment naïve for any of the following: a. GnRH analogues b. Androgen receptor antagonists, or c. Androgen synthesis inhibitors (e.g. abiraterone)
* Agrees to practice contraception during the entire study treatment period and for 3 months after the last dose of IMP is administered: a. Either by using double barrier contraception, b. or, is truly sexually abstinent, when this is in line with the preferred and usual lifestyle of the participant
* Has provided written (personally signed and dated) informed consent before completing any study-related procedure, which means any assessment or evaluation that would not have formed a part of his normal medical care

Exclusion Criteria:

* Has abnormal screening and/or baseline laboratory values that suggest a clinically significant underlying disease, or the following laboratory values: a. Liver function test (aspartate aminotransferase [ASAT/SGOT], alanine aminotransferase [ALAT/SGPT]), or total bilirubin exceeding twice the upper limit of the normal (ULN) range b. Creatinine twice the ULN range c. Uncontrolled diabetes (HbA1c >7.5%) or previously undiagnosed diabetes mellitus with HbA1c >6.5%
* Has any contraindication to the use of teverelix TFA
* Has life expectancy of less than 1 year
* Has T levels <2.0 ng/mL at screening
* Has a medical history of bilateral orchidectomy
* Using any of the following prohibited treatments: a. Within 25 weeks prior to screening: dutasteride b. Within 12 weeks prior to screening: finasteride c. Current use of any of the following: i. Anti-androgen therapy, including T replacement therapy and 5α-reductase inhibitor treatment etc. ii. GnRH analogues, androgen receptor antagonists iii. Androgen synthesis inhibitors (e.g. abiraterone) iv. Any other medication or herbal product that may affect hormone levels and might, therefore, confound interpretation of the study results (e.g. St. John's wort)
* Has neurological disease, psychiatric disease, drug or alcohol abuse, which could interfere with the participant's proper compliance
* Has a history of myocardial infarction, unstable symptomatic ischaemic heart disease, any ongoing cardiac arrhythmias of grade >2 (chronic stable atrial fibrillation on stable anticoagulant therapy is allowed), thromboembolic events (e.g. deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other significant cardiac condition (e.g. pericardial effusion, restrictive cardiomyopathy) within 6 months before screening
* Has congenital long QT syndrome or ECG abnormalities at screening of: a. Q-wave infarction, unless identified ≥6 months before screening b. Fridericia corrected QT interval (QTcF interval) >480 msec. If QTcF is prolonged in a participant with a pacemaker, the participant may be enrolled in the study upon discussion with the project clinician c. If the QTcF interval is 450-480 msec, inclusive, in a participant with current use of medications with known effects on QT interval, the participant may be enrolled in the study following discussion with the Medical Lead
* Has known or suspected severe renal impairment
* Has a medical history of diagnosis of, or treatment for, another malignancy within 2 years before the first dose of IMP, or previous diagnosis of another malignancy with evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Is currently using Class IA (e.g. quinidine, procainamide) or Class III (e.g. amiodarone, sotalol) antiarrhythmic medications
* Has uncontrolled hypertension despite appropriate medical therapy (sitting BP of >180 millimetres of mercury [mmHg] systolic and >95 mmHg diastolic at 2 separate measurements taken no more than 60 minutes apart during the screening visit). Participants with isolated systolic BP measurements >180 mmHg may be rescreened. Participants with isolated systolic BP measurements 141 to 180 mmHg or isolated diastolic BP measurements ≥95 mmHg, although eligible, should be referred for further management of hypertension if indicated
* Has known, previously diagnosed human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C, life-threatening illness unrelated to prostate cancer, or any serious medical condition that could, in the investigator's opinion, potentially interfere with participation in this study. Specific screening for chronic viral illness is at the discretion of the site and/or local Institutional Review Board (IRB)
* Has been exposed to another investigational drug within the 3 months prior to screening
* Has anticipated non-availability for study visits/procedures
* Plans to undergo surgery during the study period
* Known presence of hepatic metastases

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albertas Ulys, MD, Principal Investigator — National Cancer Institute, Vilnius, Lithuania
Locations (4):
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda University Hospital, Klaipėda
  - National Cancer Institute, Vilnius
  - Vilnius University Hospital Santaros Clinic, Vilnius

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Started | 9 | 41
Completed | 5 | 32
Not Completed | 4 | 9

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly | Total
Number analyzed (Participants) | 9 | 41 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 9 | 11
  >=65 years | 7 | 32 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (5.12) | 69.0 (7.33) | 69.0 (6.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 41 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 9 | 41 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  Lithuania | 9 | 41 | 50

OUTCOME MEASURES:

1. Primary Outcome: Testosterone (T) Levels (Castrate) at Week 4
Description: Proportion of participants achieving castration level with serum T <0.5 ng/mL at Day 28.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 9 | 41
Participants | 5 | 39

2. Secondary Outcome: Testosterone (T) Levels (0.2 ng/mL) at Week 4
Description: Proportion of participants achieving castration level with serum T <0.2 ng/mL at Day 28
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 9 | 41
Participants | 2 | 32

3. Secondary Outcome: Testosterone (T) Levels (Castrate) at Week 6
Description: Proportion of participants achieving castration level with serum T <0.5 ng/mL at Day 42
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 9 | 41
Participants | 4 | 33

4. Secondary Outcome: Testosterone (T) Levels (0.2 ng/mL) at Week 6
Description: Proportion of participants achieving profound castration level (0.2 ng/mL) with serum T <0.5 ng/mL at Day 42
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 9 | 41
Participants | 1 | 26

5. Secondary Outcome: Testosterone Levels (Castrate) at Week 24
Description: Proportion of participants achieving a T castration rate over 168 days of treatment period
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 9 | 41
Participants | 3 | 27

6. Secondary Outcome: Testosterone Levels (0.2 ng/mL) at Week 24
Description: Proportion of participants achieving profound castration rate (<0.2 ng/mL) over 168 days of treatment period
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 9 | 41
Participants | 0 | 17

7. Secondary Outcome: Time to Achieve Castrate Levels of Testosterone (T)
Description: Mean time to T levels falling below castration level (<0.5 ng/mL) for the first time
Time Frame: 4 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
days | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 3.0]

8. Secondary Outcome: Time to Escape Castrate Levels of Testosterone (T)
Description: Mean time to (first) overstep of T castration level after achieving castration
Time Frame: Approximately 30 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
days | 2.5 [1.0 to 123.0] | 215.0 [42.0 to 236.0]

9. Secondary Outcome: Luteinizing Hormone (LH) Levels (Castrate) at Week 4
Description: Proportion of participants achieving castration level for LH (LH <1.1 U/L) at Day 28
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 9 | 41
Participants | 5 | 38

10. Secondary Outcome: Luteinizing Hormone (LH) Levels (Castrate) at Week 24
Description: Proportion of participants with effective LH castration rate over 168 days of treatment period
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 9 | 41
Participants | 2 | 22

11. Secondary Outcome: Time to Achieve Castrate Levels of Luteinizing Hormone (LH)
Description: Mean time to LH levels falling below castration level (LH <1.1 U/L) for the first time
Time Frame: 4 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
days | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

12. Secondary Outcome: Time to Escape Castrate Levels of Luteinizing Hormone (LH)
Description: Mean time to (first) overstep of LH castration level after achieving castration
Time Frame: 24 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
days | 4.5 [2.0 to 83.0] | 8.5 [2.0 to 42.0]

13. Secondary Outcome: Change in Testosterone Levels Over Time (Change From Baseline at Day 168)
Description: The change in testosterone levels over time (Change from Baseline at Day 168)
Time Frame: 24 weeks
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
nmol/L | -16.68 (5.43) | -20.26 (7.37)

14. Secondary Outcome: Change in LH Levels Over Time
Description: The change in LH levels over time
Time Frame: 24 weeks
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
IU/L | -69.8825 (22.99177) | -83.3425 (26.87486)

15. Secondary Outcome: Change in FSH Levels Over Time
Description: The change in FSH levels over time
Time Frame: 24 weeks
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
IU/L | -71.8909 (12.83868) | -82.3272 (12.67620)

16. Secondary Outcome: Area Under the Concentration Time-curve From Time Zero up to the Last Quantifiable Concentration at Time Point t (AUC0-t)
Description: Area under the concentration time-curve from time zero up to the last quantifiable concentration at time point t (Ct), calculated using the linear up/log down trapezoidal rule.
Time Frame: 24 weeks
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 39
h*ng/mL | 16007 [10118.4 to 25316.4] | 27511 [23235.6 to 32573.7]

17. Secondary Outcome: Area Under the Concentration Time-curve From Time Zero up to the Concentration at Time Point t1 After Which the Concentrations Start to Rise Again Towards a Second Peak (AUC0-t1)
Description: Area under the concentration time-curve from time zero up to the concentration at time point t1 after which the concentrations start to rise again towards a second peak, calculated using the linear up/log down trapezoidal rule. t1 will be determined after review of the concentration-time profiles (immediate release component of total observed AUC).
Time Frame: 24 weeks
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 39
h*ng/mL | 1324.3 [928.2 to 1892.1] | 1759.3 [1581 to 1958.4]

18. Secondary Outcome: Maximum Observed Plasma Teverelix Concentration After Administration (Cmax)
Description: The maximum observed plasma teverelix concentration after administration (Cmax)
Time Frame: 24 weeks
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 39
ng/mL | 38.22 [30.6 to 45.9] | 53.1 [45.9 to 56.1]

19. Secondary Outcome: Maximum Observed Concentration After Administration From Zero up to Time Point t1 (Cmax,0-t1)
Description: The maximum observed concentration after administration from zero up to time point t1 (Cmax,0-t1)
Time Frame: 24 weeks
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 39
ng/mL | 38.22 [30.6 to 45.9] | 53.1 [45.9 to 56.1]

20. Secondary Outcome: Maximum Observed Concentration After Administration From Time Point t1 up to Time Point t (Cmax,t1-t)
Description: The maximum observed concentration after administration from time point t1 up to time point t (Cmax,t1-t)
Time Frame: 24 weeks
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
ng/mL | 16.9 [10.2 to 25.5] | 20.4 [20.4 to 25.5]

21. Secondary Outcome: Time to Reach Cmax After Dosing (Tmax)
Description: The time to reach Cmax after dosing (tmax)
Time Frame: 24 weeks
Population: Per Protocol
Measure: Median (Full Range); unit: hours
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 39
hours | 1.8 [1.0 to 2.6] | 1.5 [0.9 to 3.2]

22. Secondary Outcome: Time to Reach Cmax,0-t1 After Dosing (Tmax,0-t1)
Description: The time to reach Cmax,0-t1 after dosing (tmax,0-t1)
Time Frame: 24 weeks
Population: Per Protocol
Measure: Median (Full Range); unit: hours
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 39
hours | 1.8 [1.0 to 2.6] | 1.5 [0.9 to 3.2]

23. Secondary Outcome: Time to Reach Cmax,t1-t After Dosing (Tmax,t1-t)
Description: The time to reach Cmax,t1-t after dosing (tmax,t1-t)
Time Frame: 24 weeks
Population: Per Protocol
Measure: Median (Full Range); unit: hours
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 39
hours | 96.0 [72.0 to 333.6] | 167 [71.0 to 527.9]

24. Secondary Outcome: Apparent Terminal Elimination Rate Constant (Lambda-z)
Description: The apparent terminal elimination rate constant (lambda-z)
Time Frame: 24 weeks
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: L/h
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 39
L/h | 0 [0 to 0] | 0 [0 to 0]

25. Secondary Outcome: Apparent Terminal Plasma Half-life (t½)
Description: Apparent terminal plasma half-life, calculated as: ln 2 / lambda-z
Time Frame: 24 weeks
Population: Per Protocol
Measure: Median (Full Range); unit: hours
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 39
hours | 1380.3 [198.5 to 7827] | 1103.1 [209.7 to 4242]

26. Secondary Outcome: Area Under the Concentration Time-curve From Time Zero up to Infinity (∞)(AUC0-∞)
Description: Area under the concentration time-curve from time zero up to infinity (∞),calculated using the linear up/log down trapezoidal rule.
Time Frame: 24 weeks
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 39
h*ng/mL | 24888 [12693.9 to 48796.8] | 35794 [29952.3 to 42778.8]

27. Secondary Outcome: Prostate Specific Antigen (PSA) Reduction (≥50 Percent)
Description: Number of participants with a PSA response of ≥50 percent reduction at the Day 168 visit
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
Participants | 5 | 30

28. Secondary Outcome: PSA Response Rate at Day 28
Description: PSA response is defined as >50% decline in PSA at Day 28. PSA response rate is the number of subjects with a PSA response.
Time Frame: 24 weeks
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
Participants | 6 | 35

29. Secondary Outcome: PSA Response ≥50% at Day 168
Description: The number of subjects with a PSA response ≥50% at Day 168
Time Frame: 24 weeks
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
Participants | 5 | 30

30. Secondary Outcome: Luteinizing Hormone (LH) Mean % Reduction at Day 168
Description: Luteinizing Hormone (LH) - the mean % reduction at Day 168
Time Frame: 24 weeks
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: % of baseline value
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
% of baseline value | -69.88 (22.99) | -83.34 (26.87)

31. Secondary Outcome: Testosterone (T) Mean % Reduction at Day 168
Description: Testosterone (T) - the mean % reduction at Day 168
Time Frame: 24 weeks
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: % of baseline
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
% of baseline | -91.1 (7.02) | -95.9 (4.57)

32. Secondary Outcome: Follicle Stimulating Hormone (FSH) Mean % Reduction at Day 168
Description: Follicle Stimulating Hormone (FSH) - the mean % reduction at Day 168
Time Frame: 24 weeks
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: % of baseline
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 8 | 40
% of baseline | -71.89 (12.84) | -82.33 (12.68)

33. Secondary Outcome: Treatment-emergent Adverse Events (AEs)
Description: Number of participants with treatment-emergent AEs
Time Frame: 24 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 9 | 41
Participants | 8 | 38

34. Secondary Outcome: ECG QTcF Interval Prolongation >450 Msec at Day 28
Description: ECG QTcF Interval prolongation >450 msec at Day 28 study visit
Time Frame: 24 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 9 | 41
Participants | 1 | 3

35. Secondary Outcome: Injection Site Reactions (ISRs)
Description: Number of participants with ISRs at each visit during the 168 days treatment period
Time Frame: 24 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
Number analyzed (Participants) | 9 | 41
Participants | 5 | 26

ADVERSE EVENTS:
Time Frame: Until 30 days after last injection of study drug
Arm/Group | Teverelix TFA 120 mg 6-weekly | Teverelix TFA 180 mg 6-weekly
All-Cause Mortality (participants affected / at risk) | 0/9 | 1/41
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/41
Other Adverse Events (participants affected / at risk) | 8/9 | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teverelix TFA 120 mg 6-weekly (N=9) | Teverelix TFA 180 mg 6-weekly (N=41)
Left Carotid Artery Stenosis (Vascular disorders) | 1 (1) | 0 (0) — The patient was hospitalized for planned treatment due to Left Carotid Artery Stenosis (CTCAE Grade 3).
benign pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Study drug was discontinued as exclusion criterion was met.
cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) — A 75 year old, in Group 2, had a cardiac arrest on Day 196 during follow-up period of the study and subsequently died.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teverelix TFA 120 mg 6-weekly (N=9) | Teverelix TFA 180 mg 6-weekly (N=41)
Injection site induration (General disorders) | 7 (7) | 30 (30)
Injection site erythema (General disorders) | 6 (6) | 29 (29)
Injection site swelling (General disorders) | 3 (3) | 5 (5)
Induration (General disorders) | 0 (0) | 3 (3)
Injection site pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 4 (4) | 17 (17)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 5 (5)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 4 (4)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nephrostomy (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT04693507/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT04693507/SAP_001.pdf